CLINICAL TRIAL: NCT00353925
Title: Genetic Analysis of African-American Hypertensives
Brief Title: Genetic Analysis of African-Americans With High Blood Pressure
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 000003; 00-H-0003
Record Dates: First submitted 2006-07-18; First posted 2006-07-19 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2007-12-10

CONDITIONS: Hypertension
Keywords: Hypertrophy; LVH; Cardiac; Blood Pressure; Papillary Muscle
MeSH Terms: conditions — Hypertension; Hypertrophy

SUMMARY:
The purpose of this study is to learn if kinase, a protein found in the heart, contributes to thickening of the heart muscle in people with high blood pressure.

A protein called myosin causes the heart to contract and relax. It is thought that kinase changes myosin to make it work better at different heart rates. This study will try to determine if, in some people with high blood pressure, the different forms of this protein cause changes in the heart. If the protein affects the size of the heart, it might be possible to use it to improve heart function after an injury, such as a heart attack.

African-Americans with high blood pressure will be eligible for this study. Current data show that of almost 900 multi-ethnic individuals, the particular form of kinase under study in this project is found exclusively in the African-American population. Study participants will have two tubes of blood drawn for DNA testing to determine what form of kinase is present. An electrocardiogram will also be done if a recent one is not available. Some people may also have an echocardiogram, an ultrasound test to image the heart.

DETAILED DESCRIPTION:
Genetic and in vitro mechanical studies in our laboratory have suggested that the perturbations in the phosphorylation of the cardiac myosin regulatory light chain (RLC) can modulate cardiac function and produce a compensatory hypertrophic response. We have cloned a novel human cardiac kinase (MLCK) that targets the cardiac RLC and identified a common allele unique to the African-American population. The purpose of this protocol is to evaluate a large group of African-American individuals with hypertension and/or cardiac disease, a portion of who will possess this allele. It is well documented that hypertensive African-Americans have an increased prevalence of left ventricular hypertrophy (LVH). We expect that, in this population of hypertensive individuals, we will find an increased left ventricular mass in individuals who are heterozygous or homozygous for this kinase allele.

In this study, patients with the allele can be matched to others in the cohort without the allele and evaluated by echocardiography and cardiac MRI to evaluate cardiac function and chamber size. In addition, metabolic stress testing will be performed to assess the implications of this allele on clinical performance. Another group of 75 Afro-Americans with dilated cardiomyopathy will be referred from local heart failure clinics and evaluated in a similar fashion. Allele prevalence and associated cardiac findings will also be compared with hypertensive patients matched for age and gender. In a parallel experiment, mice over-expressing this kinase, are being generated and will provide us with tissue samples with which to pursue the biophysical basis of the mechanical changes in muscle function.

ELIGIBILITY:
* INCLUSION CRITERIA:

Inclusion Criteria (Main Cohort):

Afro-American patients with a history of hypertension

Age greater than or equal to 21 years old

Presence of the kinase allele (homo or heterozygous)

Ability to give informed consent.

Inclusion Criteria (Myopathy Cohort):

All of the above as well as:

Left ventricular ejection fraction of less than 35% by any imaging technique.

EXCLUSION CRITERIA

For subjects with Kinase Allele:

There will be no exclusion criteria. Patients will be evaluated even if they are only able to participate in part of the study.

For Subjects without the kinase allele and Myopathy Cohort:

History of myocardial infarction

History of significant valve disease

History of primary hyperthropic or infiltrative cardiomyopathy

History of rheumatic heart disease

Chronic atrial arrhythmia, bundle branch block intraventricular conduction defect or definite myocardial infarction on EKG

Inability to perform a metabolic stress test

Inability to perform a cMRI

Poor echocardiographic windows precluding accurate analysis

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000
Dates: Start 1999-10-05; Study Completion 2007-12-10

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland, Baltimore, Baltimore, Maryland, United States

REFERENCES:
- [Background] Sahn DJ, DeMaria A, Kisslo J, Weyman A. Recommendations regarding quantitation in M-mode echocardiography: results of a survey of echocardiographic measurements. Circulation. 1978 Dec;58(6):1072-83. doi: 10.1161/01.cir.58.6.1072. PMID 709763